CLINICAL TRIAL: NCT05439005
Title: Opioid Free Versus Opioid Based Anaesthesia for Free Flap Reconstruction Surgery of the Breast: A Phase III Multicentric Randomized Controlled Study.
Acronym: OFOBA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IC 2021-07
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: free flap reconstruction surgery; anaesthesia
MeSH Terms: conditions — Breast Neoplasms | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OFA group (Experimental): OFA (Opioid Free Anaesthesia) group:
  Interventions: Drug: Dexmedetomidine
- CA control group (No Intervention): CA (Conventional Anaesthesia) control group:

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine+Lidocaine
  Arms: OFA group

SUMMARY:
This study will compare morphine consumption during the first 48 hours postoperatively between the OFA group and the CA control group.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 or older.
2. Patients with a French health insurance coverage (having a French social security number).
3. Patient eligible for free flap reconstruction surgery of the breastunder general anaesthesia.
4. Patient who has given written consent to participate in accordance with the regulations.
5. Having a negative blood pregnancy test for patients of childbea ring age.

Exclusion Criteria:

1. Allergy or intolerance to any of the drugs (dexmedetomidine, remifentanil, lidocaine, propofol, dexamethasone, kétamine, ketoprofen, nefopam, paracetamol, morphine, ropivacaine, droperidol, ondansetron).
2. Known history of heart failure, arrhythmias and/or ischemic heart disease and/or severe renal insufficiency.
3. Pulse below 50bpm during anaesthesia consultation and/or under beta blocker treatment.
4. Treatment with ACEI/ARB.
5. Severe asthma.
6. Symptomatic gastric or duodenal ulcer with or without treatment.
7. Baseline systolic blood pressure < 100 mmHg.
8. Chronic preoperative pain and/or use of WHO ladder step 2 or 3 analgesics preoperatively.
9. Patient already included in another therapeutic trial evaluating an experimental molecule.
10. Persons deprived of liberty or under guardianship.
11. Patients with suspected difficulties in assessing pain on a scale.
12. Inability to undergo trial medical monitoring due to geographic, social or psychological reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient eligible for free flap reconstruction surgery of the breastunder general anaesthesia.
Enrollment: 158 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2027-06-06 (Estimated); Study Completion 2027-06-06 (Estimated)

PRIMARY OUTCOMES:
comparison of Morphine consumption in the two groups | during the first 48 hours postoperatively

SECONDARY OUTCOMES:
Assessment of vasopressor requirement and total intraoperative filling volume | end of surgery
Assessment of the state of consciousness on arrival in the PACU | on arrival in the PACU
Assessment of the incidence of PONV in the PACU, at D0, D1 and D2 | in the PACU, at D0, D1 and D2
Maximum VAS at rest and mobilization in the PACU, at D0, D1 and D2 | in the PACU, at D0, D1 and D2
Dose of morphine given in titration in the PACU (mg) | in the PACU
Number of boluses demand on PCA during the first 48 hours postoperatively | the first 48 hours postoperatively
DN3 score (Neuropathic Pain 3) on D2, D4, M1, M3 and M6 | on D2, D4, M1, M3 and M6
Length of stay in PACU (h) and length of in-hospital postoperative length of stay (D) | at discharge
Assessment of the flap failure rate (flap removal surgery) and flap micro-anastomosis re-exploration rate | at discharge
Pain management satisfaction scores (score from 0 to 10) at discharge | at discharge
Collection of serious adverse events between D0 (date of surgery) and D30 | between D0 (date of surgery) and D30
Dose of intraoperative rescue remifentanil in the OFA group (mcg) | at discharge
Morphine consumption during the first 48 hours post-operatively (mg) in each breast reconstruction subgroup (immediate and secondary); | the first 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Mary SAAD, MD, Study Director — Institut Curie Saint-Cloud
Locations (3):
- France (3):
  - Institut Curie Paris, Paris
  - Institut Curie Saint-Cloud, Saint-Cloud
  - Gustave Roussy, Cancer Campus, Grand Paris, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified data sets with interested researchers, educators or clinicians. Materials generated under the project will be disseminated in accordance with Institut Curie policies.
Time Frame: Data requests can be submitted starting 9 months after article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific reserach, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Derived] Saad-Boutry M, Carton M, Ezzili C, Savignoni A. Opioid-free versus opioid-based anaesthesia for free-flap reconstruction surgery of the breast: protocol for a phase III, multicentre, randomised controlled study. BMJ Open. 2025 Feb 17;15(2):e070021. doi: 10.1136/bmjopen-2022-070021. PMID 39961716